CLINICAL TRIAL: NCT00041015
Title: An Open-Label, Multicenter, Randomized, Phase III Study Comparing Oral Topotecan/Cisplatin Versus Etoposide/Cisplatin As Treatment For Chemotherapy-Naive Patients With Extensive Disease - Small Cell Lung
Brief Title: Combination Chemotherapy in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKF1501; CWRU-070144; SB-389; SB-SKF-104864A; SB-SKF-1501; NCI-G02-2092
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Cisplatin; Etoposide; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral topotecan plus cisplatin IV (Active Comparator): oral topotecan once daily on days 1-5 and cisplatin IV on day 5
  Interventions: Drug: cisplatin; Drug: topotecan hydrochloride
- Cisplatin IV plus etoposide IV (Experimental): Cisplatin IV on day 1 and etoposide IV over at least 30 minutes
  Interventions: Drug: cisplatin; Drug: etoposide

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
  Arms: Cisplatin IV plus etoposide IV
Drug: topotecan hydrochloride
  Arms: oral topotecan plus cisplatin IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating extensive-stage small cell lung cancer.

PURPOSE: Randomized phase III trial to compare different chemotherapy regimens in treating patients who have extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with chemotherapy-naive extensive stage small cell lung cancer treated with cisplatin and oral topotecan vs cisplatin and etoposide.
* Compare the response rates, response duration, and time to progression in patients treated with these regimens.
* Compare the tolerability of these regimens in these patients.
* Compare the patient-perceived disease status and well being in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to gender, ECOG performance status (0 vs 1 vs 2), lactate dehydrogenase (less than 1.5 times upper limit of normal (ULN) vs 1.5 times ULN or greater), and country. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral topotecan once daily on days 1-5 and cisplatin IV on day 5.
* Arm II: Patients receive cisplatin IV on day 1 and etoposide IV over at least 30 minutes on days 1-3.

Treatment in both arms repeats every 21 days for at least 4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, prior to each course, at 4 weeks after study, and then every 4 weeks for 16 weeks.

Patients are followed at 4 weeks, every 4 weeks for 16 weeks, and then every 3 months thereafter.

PROJECTED ACCRUAL: Approximately 760 patients (380 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed extensive stage small cell lung carcinoma (SCLC)
* No prior chemotherapy for SCLC OR
* No chemotherapy within 5 years of diagnosis of SCLC
* Prior radiotherapy to measurable or nonmeasurable disease field allowed provided radiotherapy was completed at least 6 weeks ago and the disease is demonstrated to be progressing
* No clinical signs or symptoms of brain and/or leptomeningeal metastases by CT scan or MRI

  * Brain and/or leptomeningeal metastases that are asymptomatic on neurologic exam are allowed provided metastases do not require corticosteroid therapy to control symptoms

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Hemoglobin at least 9.0 g/dL
* WBC at least 3,500/mm3
* Platelet count at least 100,000/mm3
* Neutrophil count at least 1,500/mm3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT and SGPT no greater than 2 times the upper limit of normal (ULN) (5 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 2 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No pre-existing renal impairment that would preclude cisplatin use

Gastrointestinal:

* No clinical evidence of any gastrointestinal (GI) conditions including:

  * Removal of a portion of the stomach
  * History of recent obstruction of the GI tract
  * GI autonomic neuropathy
  * Ulcerative colitis
  * Crohn's disease
  * Malabsorption syndrome
  * Treatment with cyclosporine that would alter absorption or GI motility
* No other conditions that would preclude absorption of oral topotecan

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 3 months prior to study, during, and for at least 1 month after study
* No active infection
* No other prior or concurrent malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or localized low-grade prostate cancer
* No other concurrent severe medical problems that would expose the patient to extreme risk or preclude study compliance
* No prior allergic reactions to compounds chemically related to study drugs
* No pre-existing hearing impairment that would preclude cisplatin use
* No overall medical condition for which study drugs would be inappropriate

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy for SCLC

Chemotherapy:

* See Disease Characteristics
* No other concurrent chemotherapy for SCLC

Endocrine therapy:

* See Disease Characteristics
* No concurrent hormonal therapy for SCLC

Radiotherapy:

* See Disease Characteristics
* At least 24 hours since prior radiotherapy with no expected bone marrow suppression
* Recovered from prior palliative radiotherapy (e.g, nausea and vomiting from radiation of the epigastrium)
* No concurrent radiotherapy for SCLC
* No concurrent radiotherapy for palliation of bone metastases or CNS lesions unless approved by the investigator

Surgery:

* At least 3 weeks since prior major surgery (a shorter period is allowed if deemed in the best interest of the patient)

Other:

* More than 30 days or 5 half-lives (whichever is longer) since prior investigational drugs
* No other concurrent investigational therapy for SCLC
* No concurrent cyclosporine
* No concurrent drugs that would preclude absorption of oral topotecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2001-09; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Levitan, MD, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States